CLINICAL TRIAL: NCT04524624
Title: A Multi-centre, Cluster Randomized Controlled Trial of an Artificial Intelligence-Based Clinical Decision Support System for Integrated Management of Patients With Acute Ischemic Stroke: The GOLDEN BRIDGE II Trial
Brief Title: An AI-Based CDSS for Integrated Management of Patients With Acute Ischemic Stroke(GOLDEN BRIDGE II)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Principal Investigator, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY 2020-016-02
Record Dates: First submitted 2020-08-07; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: acute ischemic stroke; artificial intelligence; clinical decision support system; cluster randomized controlled trial; evidence-based performance
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-based CDSS (Experimental): 1. Automatically identifying acute ischemic stroke lesions on DWI.
  2. Classification of stroke subtypes and mechanisms.
  3. Evidence-based alerts and guidelines for early stroke management.
  4. Guideline-recommended secondary stroke prevention strategies.
  Interventions: Device: AI-based CDSS
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Device: AI-based CDSS — 1. Automatically identifying acute ischemic stroke lesions on DWI.
  2. Classification of stroke subtypes and mechanisms.
  3. Evidence-based alerts and guidelines for early stroke management.
  4. Guideline-recommended secondary stroke prevention strategies.
  Arms: AI-based CDSS

SUMMARY:
This study will conduct a cluster randomized controlled trial to evaluate the impact of an artificial intelligence-based clinical decision support system for the integrated management of patients with acute ischemic stroke on the adherence to guideline-based therapies and the incidence of new clinical vascular events.

DETAILED DESCRIPTION:
Artificial intelligence (AI) and clinical decision support system (CDSS) have demonstrated great progress in the diagnosis and treatment of cerebrovascular diseases.CDSS can use computer technology to simulate and extend expert knowledge and empirical evidence in a timely and efficient manner. The combination of AI and CDSS is a potential solution to the shortage of medical resources and can improve the quality of and promote the standardization of medical services. At intervention sites, neurologists will receive support on use of the AI-based CDSS.

Aim: To evaluate the effectiveness of an AI-based CDSS for stroke management in patients with acute ischemic stroke within 7 days of symptom onset.

Intervention: An AI-based CDSS for an integrated management of patients with acute ischemic stroke. The strategy includes automatically identifying acute stroke lesions and lesion patterns, automated classification of stroke subtypes and mechanisms, evidence-based alerts, and guideline-recommended secondary stroke prevention strategies.

Eighty eligible hospitals in china, stratified by hospital capacity (secondary grade or tertiary) and economic-geographical regions (eastern, central, and western), will be randomized into either the CDSS group or the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* Cluster Inclusion Criteria:

  * Secondary or tertiary hospitals with an emergency department and neurologic wards that receive patients with AIS.
  * Hospitals with available brain MRI scans (1.5T or 3.0T).
* Patient Inclusion Criteria:

  * Patients of 18 years or older.
  * Patients admitted with neurological deficit consistent with ischemic stroke within 7 days of of symptoms onset. (*Symptom onset is defined by the "last seen normal" principle)
  * Confirmation of new ischemic stroke by objective modality of CT scan and MRI (had relevant lesions on DWI).
  * Informed consent from patient or legally authorised representative (primarily spouse, parents, adult children, otherwise indicated).

Exclusion Criteria:

* Cluster Exclusion Criteria:

  * Grade-one hospitals and rural hospitals.
  * The specialized hospitals, such as women and children specialist hospital and tumor hospital.
  * Hospitals with less than 20 patients with suspected AIS per month.
* Patient Exclusion Criteria:

  * Diagnosed DWI negative stroke.
  * Diagnosed other types of cerebrovascular diseases, such as transient ischaemic attack, hemorrhagic stroke, cerebral venous sinus thrombosis, and so on.
  * Diagnosed non cerebral vascular disease, such as stroke mimic, seizures, central nervous system infections, metabolic encephalopathy, and so on.
  * Received carotid endarterectomy (CEA) and carotid angioplasty and stenting (CAS).
  * Involving in other investigational drug or device clinical trials.
  * Patients with malignant disease and life expectancy of less than 3 months or patients who are unable to complete the study for other reasons.
  * Women who are pregnant or postpartum (≤6 weeks).
  * Patients refuse to participate in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21689 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) | 3 months
  To evaluate the efficacy of AI-based CDSS in reducing the risk of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) at 3 months after initial symptom onset.

SECONDARY OUTCOMES:
Incidence rate of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) | 6, 12 months
  Incidence rate of new clinical vascular events (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) at discharge, 6,12-months after initial symptom onset.
Disability | 3, 6, 12 months
  Degree of disability (measured by the Modified Rankin Scale) at discharge, 3, 6, and 12 months
All-or-none measure of evidence-based performance measures | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Proportion of prescription of evidence-based performance measures. "All or none" measures including the evidence-based therapies: antithrombotic medication within 48 hours after symptom onset, dual antiplatelet therapy (aspirin and clopidogrel) started within 24 hours after symptom onset (NIHSS score ≤3), intensive statin therapy, antihypertensive, hypoglycemic medications, dysphagia screening, and deep vein thrombosis prophylaxis within 48 hours of admission. Discharge therapies include: antithrombotics, lipid lowering agents, anticoagulants for atrial fibrilation or flutter, antihypertensive, and hypoglycemic medications.
A composite measure score of performance measures | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The composite measure score was defined as the total number of eligible performance measures performed divided by the total number of performance measures for which a given patient was eligible.
All-cause mortality | 3, 6, 12 months
  All-cause mortality

OTHER OUTCOMES:
Moderate and severe bleeding events according to the GUSTO criteria | 3, 6, 12 months
  Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage.
All bleeding events | 3, 6, 12 months
  All bleeding events (severe/moderate bleeding and intracranial hemorrhage)
Intracranial hemorrhagic events | 3, 6, 12 months
  Intracranial hemorrhagic events
Total costs of care | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Total costs of care
Average length of stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Average length of stay
Home time | 3, 6, 12 months
  We calculated home time as total days alive and not in a hospital or skilled nursing facility.
All-cause readmission | 3, 6, 12 months
  All-cause readmission
Ischemic stroke readmission | 3, 6, 12 months
  Ischemic stroke readmission
Hemorrhagic stroke readmission | 3, 6, 12 months
  Hemorrhagic stroke readmission
Cardiovascular readmission | 3, 6, 12 months
  Cardiovascular readmission
Adverse events | 3, 6, 12 months
  Adverse events
Stratified analysis | 3, 6, 12 months
  Efficacy endpoint will also be analyzed stratified by Hospital level(secondary hospitals/tertiary hospitals), economic-geographical regions (eastern, central, and western), stroke severity (NIHSS≤3/NIHSS>3) and stroke subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian tan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Wang Y, Li Z, Zhao X, Wang C, Wang X, Wang D, Liang L, Liu L, Wang C, Li H, Shen H, Bettger J, Pan Y, Jiang Y, Yang X, Zhang C, Han X, Meng X, Yang X, Kang H, Yuan W, Fonarow GC, Peterson ED, Schwamm LH, Xian Y, Wang Y; GOLDEN BRIDGE-AIS Investigators. Effect of a Multifaceted Quality Improvement Intervention on Hospital Personnel Adherence to Performance Measures in Patients With Acute Ischemic Stroke in China: A Randomized Clinical Trial. JAMA. 2018 Jul 17;320(3):245-254. doi: 10.1001/jama.2018.8802. PMID 29959443
- [Derived] Li Z, Zhang X, Ding L, Jing J, Gu HQ, Jiang Y, Meng X, Du C, Wang C, Wang M, Xu M, Zhang Y, Hu M, Li H, Gong X, Dong K, Zhao X, Wang Y, Liu L, Xian Y, Peterson E, Fonarow GC, Schwamm LH, Wang Y. Rationale and design of the GOLDEN BRIDGE II: a cluster-randomised multifaceted intervention trial of an artificial intelligence-based cerebrovascular disease clinical decision support system to improve stroke outcomes and care quality in China. Stroke Vasc Neurol. 2024 Dec 30;9(6):723-729. doi: 10.1136/svn-2023-002411. PMID 37699726